CLINICAL TRIAL: NCT06328114
Title: Functional Magnetic Resonance Imaging (fMRI)-Guided Individualized Transcranial Magnetic Stimulation (TMS) for Cervical Dystonia
Brief Title: Accelerating TMS for Cervical Dystonia
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: American Academy of Neurology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00114549
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Isolated Cervical Dystonia
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Single-arm crossover study design with subjects receiving TMS at two different intensities
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The TMS intensity delivered at each TMS visit will be masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- sham TMS (Sham Comparator): Participants receive sham TMS
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)
- TMS to primary somatosensory cortex (Active Comparator): Participants received TMS sessions at primary somatosensory cortex
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (TMS) — Participants will experience two accelerated transcranial magnetic stimulation (TMS) sessions, with 12 week (three-months) gap between each session.

SUMMARY:
This study aims to investigate the impact of accelerated transcranial magnetic stimulation (TMS) on brain function and behavior in patients with focal cervical dystonia. Previous research demonstrated that individualized TMS improved writing behavior in focal hand dystonia after one session. In this study, we aim to expand the application on TMS on focal cervical dystonia. The current study administers four TMS sessions in a day. The research involves 9 in-person visits. The effect of TMS will be assessed using functional MRI brain scans and behavioral measurements. The risk of TMS includes seizures; the potential risk of seizures from TMS is mitigated through careful screening, adhering to safety guidelines. The study's main benefit is enhancing dystonic behavior and deepening the understanding of brain changes caused by TMS in cervical dystonia, paving the way for further advancements in clinical therapy for this condition.

DETAILED DESCRIPTION:
The primary aim of this research is to investigate the impact of transcranial magnetic stimulation (TMS) on both brain function and behavioral outcomes among individuals with cervical dystonia. A previous TMS study carried out by our team revealed that the application of TMS using a personalized brain targeting approach in focal hand dystonia resulted in improved measures of writing disfluency and changes in the motor network. This study seeks to expand these promising findings to individuals with cervical dystonia. Subjects in the study will receive four TMS sessions in a single day with a protocol referred to as "accelerated TMS." The investigation will consist of a total of 9 in-person appointments. Participants with cervical dystonia will receive accelerated TMS during two in-person visits. Following each TMS session, participants will evaluate changes in brain function using function MRI and behavior using a behavior assay. The principal risk associated with TMS is the possibility of inducing a seizure. However, this study will strictly adhere to safety guidelines, utilizing TMS levels that have not previously been linked to seizures in properly screened individuals. The dosages of TMS proposed for use in this study have not caused seizures in healthy volunteers. To further mitigate the risk of seizures, potential subjects will undergo medical screening for any known factors that could predispose them to seizures. The primary advantage of this study is that it may improve neck movement behavior in patients with cervical dystonia, while also advancing our understanding in brain function before and after TMS intervention. The discoveries stemming from this investigation will pave the way for future research endeavors aimed at advancing brain stimulation as a viable clinical therapy for cervical dystonia.

ELIGIBILITY:
Inclusion Criteria:

* 18yrs and older
* Diagnosed with isolated cervical dystonia by Neurologist
* Must be able to sign an informed consent
* Must be literate

Exclusion Criteria:

* Other neurological movement disorders diagnoses including other types of dystonia, Parkinsonism, or essential tremor
* History of seizure disorder
* Concomitant medications known to decrease seizure threshold
* Illicit drug use
* No TMS therapy for another indication within one month of this research study
* Botulinum toxin injections within 3 months of the research study
* Medications used for symptom treatment of dystonia including anticholinergic, benzodiazepines, and muscle relaxants among others within one month of the study
* No physical or occupational therapy of the neck within one month of the study
* Any contraindications to MRI or TMS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2029-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in Neck Angles as Measured by Neck Sensor Device | Baseline, approximately 7 months (visit 9)
  Mixed modeling will be used to compare the degree of neck angle movements between active TMS, sham TMS, and baseline visits.

SECONDARY OUTCOMES:
Changes in Brain Activity (bold activity) on Functional Magnetic Resonance Imaging (fMRI) | Baseline (visit 1) to approximately 4 weeks (visit 7)
  The investigators will conduct a region of interest analysis in the motor network of the brain to calculate changes of fMRI bold activity after each TMS session.
Changes in Brain Activity (functional connectivity) on Functional Magnetic Resonance Imaging (fMRI) | Baseline (visit 1) to approximately 4 weeks (visit 7)
  The investigators will conduct a region of interest analysis in the motor network of the brain to calculate changes of fMRI functional connectivity after each TMS session.
Behavioral Response After Deep Brain Stimulation (DBS), as measured by Neck Angles | Approximately 6 weeks post-DBS (visit 8), approximately 7 months (visit 9)
  If participants undergo DBS, the investigators will collect neck angles over time post-DBS and correlate with the subject's neck angles over time post-TMS.

CONTACTS AND LOCATIONS:
Overall Officials: Noreen Bukhari-Parlakturk, MD PhD, Principal Investigator — Duke Health
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Noreen Bukhari-Parlakturk, Patrick Mulcahey, Michael Lutz, Rabia Ghazi, Ziping Huang, Moritz Dannhauer, Zeynep Simsek, Skylar Groves, Mikaela Lipp, Michael Fei, Tiffany Tran, Eleanor Wood, Lysianne Beynel, Burton Scott, Pichet Termsarasab, Chris Petty, Hussein R Al-Khalidi, James Voyvodic, Lawrence G. Appelbaum, Simon Davis, Andrew Michael, Angel Peterchev, Nicole Calakos. "Functional MRI-guided individualized TMS modifies motor network and reduces writing dysfluency in Focal Hand Dystonia." Human Brain Mapping Conference. Montreal, Canada. July 22-26, 2023. virtual poster presentation.
- [Background] Noreen Bukhari-Parlakturk, Patrick Mulcahey, Michael Lutz, Rabia Ghazi, Ziping Huang, Moritz Dannhauer, Zeynep Simsek, Skylar Groves, Mikaela Lipp, Michael Fei, Tiffany Tran, Eleanor Wood, Lysianne Beynel, Burton Scott, Pichet Termsarasab, Chris Petty, Hussein R Al-Khalidi, James Voyvodic, Lawrence G. Appelbaum, Simon Davis, Andrew Michael, Angel Peterchev, Nicole Calakos. "Functional MRI-guided individualized TMS modifies motor network and reduces writing dysfluency in Focal Hand Dystonia." Samuel Belzberg 6th International Dystonia Symposium. Dublin, Ireland. June 1-3, 2023. poster presentation.
- [Background] Bukhari-Parlakturk N, Lutz MW, Al-Khalidi HR, Unnithan S, Wang JE, Scott B, Termsarasab P, Appelbaum LG, Calakos N. Suitability of Automated Writing Measures for Clinical Trial Outcome in Writer's Cramp. Mov Disord. 2023 Jan;38(1):123-132. doi: 10.1002/mds.29237. Epub 2022 Oct 13. PMID 36226903
- [Background] Dannhauer M, Huang Z, Beynel L, Wood E, Bukhari-Parlakturk N, Peterchev AV. TAP: targeting and analysis pipeline for optimization and verification of coil placement in transcranial magnetic stimulation. J Neural Eng. 2022 Apr 21;19(2):10.1088/1741-2552/ac63a4. doi: 10.1088/1741-2552/ac63a4. PMID 35377345